CLINICAL TRIAL: NCT04285203
Title: Living Donation and Kidney Transplantation Information Made Easy (KIDNEYTIME) With Animated Video Education
Brief Title: Living Donation and Kidney Transplantation Information
Acronym: KIDNEYTIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Liise Kayler, Clinical Professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00002771
Record Dates: First submitted 2020-02-10; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Educational Video (Experimental): Participants were exposed to 2 educational videos in addition to standard of care education.
  Interventions: Other: Educational Video Intervention
- Standard of Care (No Intervention): Participants received standard of care education.

INTERVENTIONS:
Other: Educational Video Intervention — Educational videos
  Arms: Educational Video

SUMMARY:
The purpose of this study is to increase awareness and knowledge regarding the risks and benefits of kidney transplantation and living donation amongst patients seeking kidney transplantation and their family and friends in Buffalo, New York.

DETAILED DESCRIPTION:
This prospective randomized parallel controlled trial of kidney transplant candidates receiving and educational intervention and standard of care education versus standard of care education only to improve informed decision making about kidney offers.

ELIGIBILITY:
Inclusion Criteria:

* be 18 years or older,
* understand and read English (or have a support person that helps them)
* have acceptable vision to watch videos
* be able to give consent

Exclusion Criteria:

* incarcerated
* involved in the former modeling phase of animation development.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Change in knowledge | Baseline and immediately post exposure
  Assessed by knowledge survey pre and post exposure.
Change in attitude about kidney offers | Baseline and immediately post exposure
  Assessed by attitude survey pre and post exposure.

SECONDARY OUTCOMES:
Change in subjective decisional self-efficacy | Baseline and immediately post exposure
  Assessed by self-efficacy survey pre and post exposure.
Participation and decision making | 1 day (During standard of care education at time of clinic visit)
  Number of questions and value statements in regards to organ offers.

CONTACTS AND LOCATIONS:
Overall Officials: Liise Kayler, MD, Principal Investigator — University at Buffalo
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No